CLINICAL TRIAL: NCT07241832
Title: Multifaceted Assessment of Patients With Wilson's Disease in a Low-Resource Setting in Upper Egypt: Service Integration, Psychosocial Burden, Dietary Practices, and the Geo-Spatial Disease Map
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mostafa Ahmed Hassan, residant doctor at Assiut university hospital, Assiut University
Other Study IDs: Wilson's Disease in Upper Egy
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Wilson's Disease
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: Patients aged 12 years and older with a confirmed diagnosis of Wilson's Disease based on clinical, biochemical, radiological, slit-lap examination and genetic criteria, who are on regular follow up at Assiut Liver Center, and the Specialized Wilson's Disease Clinic
  Interventions: Behavioral: KAB-pB Scores

INTERVENTIONS:
Behavioral: KAB-pB Scores — KAB-pB Scores: Quantitative measurements of Knowledge, Attitudes, Behaviors, and perceived Barriers among patients and caregivers, derived from the structured questionnaire

SUMMARY:
Wilson's disease (WD) is a rare autosomal recessive disorder of copper metabolism, caused by mutations in the *ATP7B* gene, leading to impaired copper metabolism and toxic accumulation in many organs including the liver, brain, and cornea with subsequent hepatic and neuropsychiatric manifestations (Członkowska et al., 2018). Early diagnosis and adherence to lifelong dietary restrictions and chelation therapy are critical to prevent irreversible damage (Wang et al., 2017). WD is one of the few inborn metabolic diseases that can be successfully treated, and its complications can be prevented especially if diagnosed early and managed properly (Członkowska et al., 2018). However, in low-resource settings, patients often face barriers such as delayed diagnosis, poor awareness, limited access to care, and financial constraints (Miloh et al., 2018).

The long-term nature of the disease, possibility of debilitating symptoms, requirement of life-long and daily oral intake of medicines, life-long avoidance of copper-rich foods, frequent visits to the doctor/hospitals and the need for regular investigations impact the day-to-day physical and emotional functioning of these patients, their social lives and interpersonal relationships (Unavane et al., 2022). WD affects the quality of life of not only the patients but also their families, and the impact on patients with neuro-WD is worse than that of patients with hepatic disease (Unavane et al., 2022).

Despite treatment being occasionally available, patient adherence remains suboptimal due to a range of psychosocial, geographic, behavioral, and economic barriers (Członkowska et al., 2018). Numerous studies suggest that concordance with drug therapy including compliance (taking the prescribed dose), persistence (continuing treatment over time), and adherence (following timing and dietary instructions for medication intake (Cramer et al., 2008; Masełbas et al., 2010) is particularly poor among individuals with chronic illnesses. These challenges, which also affect patients' families, significantly hinder treatment outcomes (Masełbas et al., 2010). There is a paucity of research exploring these dimensions in low- or medium-income countries, particularly in the Middle East and North Africa (MENA) region.

Despite the clinical importance of WD, there is a significant research gap in understanding the lived experiences of Upper Egyptian patients and their families. Specifically, there is limited data on knowledge, attitudes, behaviors and perceived barriers (KAB-pB) related to WD, which are essential for effective disease management and public health interventions. Health literacy and cultural beliefs often shape how patients perceive their illness, adhere to treatment, and engage with healthcare providers. In Upper Egypt, where educational and socioeconomic disparities persist, assessing KAB-B can illuminate barriers to care and inform targeted educational strategies. Moreover, caregiver burden, which is often overlooked in chronic disease research, plays a pivotal role in patient outcomes and deserves focused attention (Adelman et al., 2014; Albani et al., 2024; Macharia et al., 2023).

Geographic access to care is another pressing concern. Patients from remote areas must travel long distances to reach the WD specialized centers facing high transportation costs, unreliable transit options, and logistical challenges that can delay diagnosis and treatment (Mseke et al., 2024). Mapping the geographic distribution of patients and their travel patterns will provide critical insights into healthcare inequities and support the development of decentralized or mobile care models. Additionally, for genetic disease like WD, geographic distribution gives insights into disease clustering of foci of mutations or social behaviors like increased consanguinity (Ferenci, 2006; Gomes & Dedoussis, 2016). These findings can guide policymakers in designing more equitable healthcare systems that accommodate the needs of rare disease populations.

Dietary management is central to WD treatment, as patients must avoid copper-rich foods such as legumes (like peas, lentils, barley, millet, wheat, bran, and fava beans), nuts, fresh sweet potatoes, in addition to chocolate shellfish, liver, and commercially dried fruits (Li et al., 2022). It is well-known that traditional Egyptian diets - especially in rural communities - often include the above legumes due to cultural preferences and economic constraints. Therefore, understanding how patients navigate these dietary restrictions within their cultural and financial realities is essential for crafting practical, culturally sensitive nutritional guidelines (Nemec, 2020). Additionally, the psychosocial burden of WD including stigma, emotional distress, and coping mechanisms remains underexplored in Upper Egypt. Studies from other contexts suggest that chronic neurological and psychiatric manifestations include depression, personality changes, and cognitive

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 12 years and older with a confirmed diagnosis of Wilson's Disease based on clinical, biochemical, radiological, slit-lap examination and genetic criteria, who are on regular follow up at Assiut Liver Center, and the Specialized Wilson's Disease Clinic.
* Patients who are clinically stable and able to participate in interviews or complete surveys.

Exclusion Criteria:

* Patients experiencing acute hepatic or neurological decompensation at the time of recruitment.
* Individuals with cognitive impairments that preclude informed consent or meaningful participation.
* Patients or caregivers who refuse to provide consent.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged 12 years and older with a confirmed diagnosis of Wilson's Disease based on clinical, biochemical, radiological, slit-lap examination and genetic criteria, who are on regular follow up at Assiut Liver Center, and the Specialized Wilson's Disease Clinic
Sampling Method: Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Dietary Adherence Index: | baseline
  Dietary Adherence Index: A composite score based on the Dietary Practices Survey, reflecting the level of adherence to copper-restricted diets and the affordability challenges faced